CLINICAL TRIAL: NCT06568796
Title: Comparison of the Effects of Trigger Point Ischemic Compression Massage and Focused Extracarporeal Shock Wave Therapy on Pain Level, Muscle Strength, Joint Range of Motion, Functionality and Quality of Life in Patients With Lateral Epicondylitis: a Randomized Controlled Trial
Brief Title: Comparison of the Effects of Trigger Point Ischemic Compression Massage and Focused Extracorporeal Shoch Wave Therapy of the Patients With Lateral Epicondylitis: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Bihter Aslanyurek, Associate Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-117
Record Dates: First submitted 2024-08-12; First posted 2024-08-23 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; trigger points ıschemıc compressıon massage; focus eswt
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Focused Ekstracorporeal Shoch Wave Theraphy and Exercise (Experimental): Individuals will be administered focused ekstracorporeal shoch wave theraphy 1 day a week for 4 weeks. Individuals will exercise every day
  Interventions: Other: randomize controlled study
- Trigger Point Ischemic Compression Massage and Exercise (Experimental): Individuals will receive trigger point ischemic compression massage 2 days a week for 4 weeks. Individuals will exercise every day
  Interventions: Other: randomize controlled study
- Exercise (No Intervention): Individuals will only exercise every day.

INTERVENTIONS:
Other: randomize controlled study — eswt treatment
  Arms: Focused Ekstracorporeal Shoch Wave Theraphy and Exercise; Trigger Point Ischemic Compression Massage and Exercise

SUMMARY:
To compare the effects of Trigger Point Ischaemic Compression Massage (TPICM) and Focused Extracarporeal Shock Wave Therapy (focused ESWT) on pain level, muscle strength, Joint range of motion, functionality and quality of life in patients with lateral epicondylitis (LE) in a randomised controlled trial.

DETAILED DESCRIPTION:
The study was planned to include at least 66 patients who presented to the sports medicine clinic of Gülhane Training and Research Hospital with lateral epicondyle pain for at least 2 months, were diagnosed with lateral epicondylitis and verbally and in writing declared that they were willing to participate in the study.

Patients participating in the study;

1. assessment of pain intensity with visual analog scale (VAS)
2. Evaluation of hand grip strength with jamar hand dynamometer
3. Isokinetic muscle strength assessment of wrist muscles with biodex isokinetic system 3
4. assessment of wrist range of motion with a manual goniometer
5. Function assessment with PRTEE-T
6. DASH questionnaire
7. SF-36 quality of life assessment will be performed before and after treatment.

inclusion criteria

1. Male and female individuals aged 18-60 years
2. being diagnosed with lateral epicondilitis
3. volunteering to participate in the study

exclusion criteria from eswt treatment

1. non-cooperation
2. presence of systemic and metabolic diseases
3. malignancy, osteoporosis, fracture, blood clotting disorder, pacemaker, infection
4. pregnancy
5. utilization of another treatment for lateral epicondylitis during the study period
6. previous invasive treatment with steroids for lateral epicondylitis
7. any treatment for lateral epicondylitis in the last 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Male and female individuals between the ages of 18-60
2. being diagnosed with lateral epicondylitis
3. volunteering to participate in the study

Exclusion Criteria:

1. non-cooperation
2. presence of systemic and metabolic diseases
3. malignancy, osteoporosis, fracture, blood clotting disorder, pacemaker, infection
4. pregnancy
5. utilization of another treatment for lateral epicondylitis during the study period
6. previous invasive treatment with steroids for lateral epicondylitis
7. any treatment for lateral epicondylitis in the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
grip strenght asessment with jamar hand dynamometer | baseline-up to 4 weeks
  It will be grip strength assessment with jamar hand dynamometer
muscle strenght asessment with isocinetic system | baseline-up to 4 weeks
  It will be elbow flexor and extansor muscle strength asessment with isocinetic system
range of motion asessment with universal goniometer | baseline-up to 4 weeks
  It will be elbow range of motion asessment with universal goniometer
assessment of quality of life with quality of life questionnaire | baseline-up to 4 weeks
  It will be asessment of quality of life with life questionnaire
pain level asessment with visual analog scale | baseline-up to 4 weeks
  It will be asessment of pain level with visual analog scale
assessment of functionality with functionality questionnaire | baseline-up to 4 weeks
  It will be asessment of functionality with functionality questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Eğitim ve Araştırma Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided